CLINICAL TRIAL: NCT00169598
Title: Remission Evaluation Before Intensified Treatment in Lymphoma: Impact of Positron Emission Tomography (PET) Using Fluorine-18-Floro-Deoxyglucose (FDG) in the Therapeutic Prescription. Medico-Economic Randomised Study
Acronym: TEPELY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2000.232
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Lymphoma
Keywords: Lymphoma; positron emission tomography; stem cell transplantation; therapeutic impact
MeSH Terms: conditions — Lymphoma | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Procedure: positron emission tomography

SUMMARY:
This randomised study aimed at evaluating the medical and economical impact of positron emission tomography (PET) using fluorine-18-fluoro-deoxyglucose (FDG) in the therapeutic prescription in patients with Hodgkin's lymphoma or with large B and P cell non-Hodgkin's lymphoma. The median progression free survival, the costs and the quality of life are compared between two groups : Group 1: the results of conventional staging and of the PET are known before stem cell transplantation. Group 2: only the results of conventional staging before stem cell transplantation are known before stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

Age over 18, with Hodgkin's lymphoma or with large B and P cell non-Hodgkin's lymphoma, or after a first-line chemotherapy with at least a residual mass or after induction chemotherapy or at progression.

Stem cell transplantation would be programmed. Patients were required to give their written informed consent.

Exclusion Criteria:

Progressive cancer or diagnosed less than 5 years, except cancer in situ of the cervix and basocell skin carcinoma, kidney insufficiency or diabetes. Patients would not be pregnant or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2002-02

PRIMARY OUTCOMES:
The impact of positron emission tomography (PET) using fluorine-18-floro-deoxyglucose (FDG) in the therapeutic prescription in patients with Hodgkin's lymphoma or with large B and P cell non-Hodgkin's lymphoma.

SECONDARY OUTCOMES:
Median progression free survival
The positive and negative likelihood- ratios, the positive and negative predictive values
The costs
The one-year survival rates
The quality of life of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Gilles SALLES, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Gilles Salles, Lyon, France